CLINICAL TRIAL: NCT05927519
Title: Airtraq in Obese and Nonobese Men
Brief Title: Comparison of Airtraq in Class 2-3 Obese and Nonobese Men During Intubation: a Prospective Randomized Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zehra Ipek ARSLAN, Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: KAEK/10.bI.03
Record Dates: First submitted 2023-06-19; First posted 2023-07-03 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Obesity, Morbid; Intubation; Difficult or Failed; Video Laryngoscope; Men
MeSH Terms: conditions — Obesity, Morbid; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Intervention Model Description: Airtraq video laryngoscope will be used in morbid obese and non obese patients
Who Masked: Participant, Outcomes Assessor
Masking Description: the participant and the outcome assessor will not know which device was used in this trail
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- morbidly obese (Active Comparator): Class 2 (bmı >35) weight kg/height m2 and class 3 (bmı>40) obese men
  Interventions: Device: airtraq video laryngoscope
- nonobese (Placebo Comparator): bmı<30 weight kg/ height m2 men
  Interventions: Device: airtraq video laryngoscope

INTERVENTIONS:
Device: airtraq video laryngoscope — airtraq video laryngoscope will be used for intubations

SUMMARY:
Morbid obesity is a growing disease. Intubations of these patients mostly difficult. Video laryngoscopes have to be used during the intubation of these patients. The intubation of men is more complicated and difficult than obese women. There were no trials compared to the new video laryngoscopes in morbidly obese men. Patients will be divided into two groups; non-obese and klas 2-3 obese. Airtraq will be used for their intubation. The time for intubation will be the primary aim of this prospective randomized study. The insertion time, perioperative hemodynamic variables, and postoperative complications will also be recorded.

DETAILED DESCRIPTION:
Morbid obesity is a growing disease. Intubations of these patients mostly difficult. Video laryngoscopes have to be used during the intubation of these patients. The intubation of men is more complicated and difficult than obese women. There were no trials compared to the new video laryngoscopes in morbidly obese men. Patients will be divided into two groups; non-obese and klas 2-3 obese. Airtraq will be used for their intubation. The time for intubation will be the primary aim of this prospective randomized study. The insertion time, need of optimization menuvers, perioperative hemodynamic variables, and postoperative complications will also be recorded.

ELIGIBILITY:
Inclusion Criteria:> 18 age men gender elective operation requring intuabtion -

Exclusion Criteria:<18 age women emergency operation

-

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — men
Enrollment: 80 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2027-10-05 (Estimated); Study Completion 2027-10-05 (Estimated)

PRIMARY OUTCOMES:
intubation time | 50 seconds
  the intubation time will be recorded beginning the insertion of the Airtraq through the mouth still the endotracheal tube seen passing through the vocal cords

SECONDARY OUTCOMES:
insertion time | 20 seconds
  inserting the Airtraq through the mouth till the optimal glottic vizualization occurred
peroperative hemodynamic variable | 4 hours
  heart rate

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Kocaeli University Medical Faculty Hospital, Iamit
  - Kocaeli UniversityMedical Faculty, Kocaeli

IPD SHARING:
Plan to Share IPD: No